CLINICAL TRIAL: NCT00006125
Title: A Phase II Study of Sequential Doxorubicin and Topotecan (Dox/Topo) in Relapsed or Refractory Intermediate- or High-Grade Non-Hodgkin's Lymphoma (NHL)
Brief Title: Combination Chemotherapy in Treating Patients With Relapsed or Refractory Intermediate-Grade or High-Grade Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-59906; U10CA031946 (NIH); CLB-59906; CDR0000068140 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2000-08-03; First posted 2003-01-27 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Lymphoma
Keywords: recurrent grade 3 follicular lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult Burkitt lymphoma; anaplastic large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Burkitt Lymphoma; Lymphoma, Large-Cell, Anaplastic | interventions — Doxorubicin; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Doxorubicin + topotecan (Experimental): Patients receive doxorubicin IV over 5-10 minutes on day 1 and topotecan IV over 30 minutes on days 3-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression.
  Patients are followed every 6 months for 2 years and annually for the next 3 years.
  Interventions: Drug: doxorubicin hydrochloride; Drug: topotecan hydrochloride

INTERVENTIONS:
Drug: doxorubicin hydrochloride
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining doxorubicin and topotecan in treating patients who have relapsed or refractory intermediate-grade or high-grade non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate and time to progression in patients with relapsed or refractory intermediate or high grade non-Hodgkin's lymphoma treated with doxorubicin and topotecan.
* Determine the toxicity of this regimen in these patients.

OUTLINE: Patients receive doxorubicin IV over 5-10 minutes on day 1 and topotecan IV over 30 minutes on days 3-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression.

Patients are followed every 6 months for 2 years and annually for the next 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed recurrent or refractory non-Hodgkin's lymphoma of one of the following subtypes:

  * Follicular center lymphoma, grade 3
  * Diffuse large B-cell lymphoma
  * Diffuse large B-cell lymphoma, primary mediastinal B-cell lymphoma
  * Burkitt's lymphoma
  * High grade B-cell lymphoma, Burkitt-like
  * Anaplastic large cell lymphoma, CD30+ cell type
  * Anaplastic large cell lymphoma, T-cell type
  * Anaplastic large cell lymphoma, null-cell type
  * Anaplastic large cell lymphoma, Hodgkin's like
* Bidimensionally measurable disease NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin no greater than 2.0 mg/dL history of Gilbert's Disease
* AST no greater than 2.5 times upper limit of normal

Renal:

* Creatinine normal

Cardiovascular:

* LVEF at least 45% by MUGA or echocardiogram

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Greater than 3 weeks since prior chemotherapy (6 weeks since prior nitrosoureas or mitomycin)
* No greater than 96 mg/m2 mitoxantrone
* No greater than 400 mg/m2 prior doxorubicin or combined total doxorubicin and mitoxantrone
* No prior camptothecins
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy except steroids for adrenal failure or hormones given for nondisease conditions (e.g., insulin for diabetes)
* No concurrent dexamethasone or other steroidal antiemetics

Radiotherapy:

* Greater than 3 weeks since prior radiotherapy
* No concurrent radiotherapy except whole brain irradiation for documented CNS disease

Surgery:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-07; Primary Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Response rate | Up to 5 years

SECONDARY OUTCOMES:
Time to progression | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Nancy L. Bartlett, MD, Study Chair — Washington University Siteman Cancer Center
Locations (76):
- United States (75):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Memorial Regional Hospital Comprehensive Cancer Center, Hollywood, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Helen and Harry Gray Cancer Institute at Good Samaritan Medical Center, West Palm Beach, Florida
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Saint Anthony Medical Center, Rockford, Illinois
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Baptist Hospital East - Louisville, Louisville, Kentucky
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Veterans Affairs Medical Center - Baltimore, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Lakeland Medical Center - St. Joseph, Saint Joseph, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - Las Vegas, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Veterans Affairs Medical Center - Asheville, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - NorthEast Oncology Associates, Concord, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - Lenoir Memorial Hospital Cancer Center, Kinston, North Carolina
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Fargo, Fargo, North Dakota
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Lifespan: The Miriam Hospital, Providence, Rhode Island
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Green Mountain Oncology Group, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Virginia Oncology Associates - Norfolk, Norfolk, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., Roanoke, Virginia
  - St. Mary's Medical Center, Huntington, West Virginia
  - Ministry Medical Group - Northern Region, Rhinelander, Wisconsin
- University of Puerto Rico School of Medicine Medical Sciences Campus, San Juan, Puerto Rico

REFERENCES:
- [Result] Smith SM, Johnson JL, Niedzwiecki D, Eder JP, Canellos G, Cheson BD, Bartlett NL; Cancer and Leukemia Group B. Sequential doxorubicin and topotecan in relapsed/refractory aggressive non-Hodgkin's lymphoma: results of CALGB 59906. Leuk Lymphoma. 2006 Aug;47(8):1511-7. doi: 10.1080/10428190600581385. PMID 16966261
- [Result] Smith SM, Johnson JL, Niedzwiecki D, et al.: Sequential topoisomerase I (topo I) and topoisomerase II (topo II) inhibitors in relapsed/refractory aggressive NHL: results of CALGB 59906, a phase II study of doxorubicin and topotecan. [Abstract] Blood 104 (11): A-2500, 2004.